CLINICAL TRIAL: NCT06326866
Title: The Association of Blood Type Differences and Signal-Noise Ratio in TEOAE and DPAOE in Individuals With Normal Hearing
Brief Title: Otoacoustic Emissions in Different Blood Types
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Eyyup Kara, Assistant Professor, Istanbul University - Cerrahpasa
Other Study IDs: E-74555795-050.04-941208
Record Dates: First submitted 2024-03-18; First posted 2024-03-22 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Hearing Loss, Cochlear
Keywords: otoacoustic emissions; blood type
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Otoacoustic Emissions, Spontaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Individuals with A Rh (+) blood group: Individuals with normal hearing and whose blood group was previously determined as A Rh (+) will be included and Transient evoked Otoacoustic Emissions (TOAE) and Distortion Product Otoacoustic Emissions (DPOAE) will be performed.
  Interventions: Diagnostic Test: Otoacoustic emissions (non-invasive)
- Individuals with A Rh (-) blood group: Individuals with normal hearing and whose blood group was previously determined as A Rh (-) will be included and Transient evoked Otoacoustic Emissions (TOAE) and Distortion Product Otoacoustic Emissions (DPOAE) will be performed.
  Interventions: Diagnostic Test: Otoacoustic emissions (non-invasive)
- Individuals with B Rh (+) blood group: Individuals with normal hearing and whose blood group was previously determined as B Rh (+) will be included and and Transient evoked Otoacoustic Emissions (TOAE) and Distortion Product Otoacoustic Emissions (DPOAE) will be performed.
  Interventions: Diagnostic Test: Otoacoustic emissions (non-invasive)
- Individuals with B Rh (-) blood group: Individuals with normal hearing and whose blood group was previously determined as B Rh (-) will be included and and Transient evoked Otoacoustic Emissions (TOAE) and Distortion Product Otoacoustic Emissions (DPOAE) will be performed.
  Interventions: Diagnostic Test: Otoacoustic emissions (non-invasive)
- Individuals with AB Rh (+) blood group: Individuals with normal hearing and whose blood group was previously determined as AB Rh (+) will be included and and Transient evoked Otoacoustic Emissions (TOAE) and Distortion Product Otoacoustic Emissions (DPOAE) will be performed.
  Interventions: Diagnostic Test: Otoacoustic emissions (non-invasive)
- Individuals with AB Rh (-) blood group: Individuals with normal hearing and whose blood group was previously determined as AB Rh (-) will be included and and Transient evoked Otoacoustic Emissions (TOAE) and Distortion Product Otoacoustic Emissions (DPOAE) will be performed.
  Interventions: Diagnostic Test: Otoacoustic emissions (non-invasive)
- Individuals with O Rh (+) blood group: Individuals with normal hearing and whose blood group was previously determined as O Rh (+) will be included and and Transient evoked Otoacoustic Emissions (TOAE) and Distortion Product Otoacoustic Emissions (DPOAE) will be performed.
  Interventions: Diagnostic Test: Otoacoustic emissions (non-invasive)
- Individuals with O Rh (-) blood group: Individuals with normal hearing and whose blood group was previously determined as O Rh (-) will be included and and Transient evoked Otoacoustic Emissions (TOAE) and Distortion Product Otoacoustic Emissions (DPOAE) will be performed.
  Interventions: Diagnostic Test: Otoacoustic emissions (non-invasive)

INTERVENTIONS:
Diagnostic Test: Otoacoustic emissions (non-invasive) — There is no invasive intervention in the study. Individuals with predetermined blood types will be included in the study.

SUMMARY:
The objective of this study is to examine whether ABO and Rhesus (Rh) blood group systems have an association with distortion product otoacoustic emission (DPOAE) and transient otoacoustic emission (TEOAE) amplitudes with the hypothesis of blood groups may affect hearing thresholds.

DETAILED DESCRIPTION:
Many factors have a significant impact on otoacoustic emission (OAE) measurement and quality of analysis. Race, age and gender are among the non-pathological factors. To date there is clear data to demonstrate the association of blood types with OAEs. The aim of our research is to investigate the relation of different blood groups (ABO) and Rh factors on transient evoked OAE and distortion product OAE amplitudes and inner ear potentials, differences between ears and to contribute to the limited literature on cochlear hearing loss susceptibility and blood groups with the hypothesis that blood groups may be associated with hearing thresholds.

ELIGIBILITY:
Inclusion Criteria:

* not having hearing loss
* having a blood group card obtained from health institutions

Exclusion Criteria:

* not meeting inclusion criteria

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals between the ages of 18-26 with known blood type without hearing loss
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Signal to noise ratios | 1 month
  SNRs obtained for different frequencies in OAE In TEOAE, 1, 1.4, 2, 2.8, 4 kHz, in DPOAE 1, 1.4, 2, 2.8, 4, 6 kHz

CONTACTS AND LOCATIONS:
Overall Officials: Eyyup Kara, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Eyyup KARA, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No data sharing is planned.